CLINICAL TRIAL: NCT05884151
Title: Comparative Efficacy of Intralesional Tranexamic Acid and Platelets Rich Plasma in the Treatment of Melasma
Brief Title: Comparison of Intralesional Tranexamic Acid and Platelets Rich Plasma in the Treatment of Melasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr sana aslam, Principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cmh abbottabad321
Record Dates: First submitted 2023-05-16; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional tranexamic acid in the treatment of melasma (Active Comparator): Group A 30 patients treated with Intradermal Tranexamic acid injection (4mg/ml) for preparation an insulin syringe was used with a volume of 1ml containing 0.04 ml of TXA and the reminder being normal saline to ensure 4mg preparation in each insulin syringe
  Interventions: Drug: Tranexamic acid
- Intrlesional platelets rich plasma in the treatment of melasma (Active Comparator): Group B 30 patients prescribed with PRP (1ml) intra-dermally PRP was obtained manually by a two-step procedure using a centrifuge machine. First spin was performed at 1500 RPM for 10 minutes. Second spin was performed at 4000 RPM for 10 minutes. Thus, obtaining a two-part plasma. Upper two third was platelet poor plasma and was discarded. Lower one third was platelets rich plasma. Before injection applying 0.1 ml calcium chloride was added for each 1 ml of PRP to activate the platelets. PRP was injected 1 ml by using 30 G needle (insulin syringe) in each cm2 of melasma.
  Interventions: Drug: Platelets rich plasma

INTERVENTIONS:
Drug: Tranexamic acid — Group A 30 patients treated with Intradermal Tranexamic acid injection (4mg/ml) for preparation an insulin syringe was used with a volume of 1ml containing 0.04 ml of TXA and the reminder being normal saline to ensure 4mg preparation in each insulin syringe
  Arms: Intralesional tranexamic acid in the treatment of melasma
Drug: Platelets rich plasma — Group B 30 patients prescribed with PRP (1ml) intra-dermally PRP was obtained manually by a two-step procedure using a centrifuge machine. First spin was performed at 1500 RPM for 10 minutes. Second spin was performed at 4000 RPM for 10 minutes. Thus, obtaining a two-part plasma. Upper two third was platelet poor plasma and was discarded. Lower one third was platelets rich plasma. Before injection applying 0.1 ml calcium chloride was added for each 1 ml of PRP to activate the platelets. PRP was injected 1 ml by using 30 G needle (insulin syringe) in each cm2 of melasma.
  Arms: Intrlesional platelets rich plasma in the treatment of melasma

SUMMARY:
ABSTRACT Objective: To study the efficacy while comparing Intralesional tranexamic acid Vs Platelets rich plasma (PRP) in treatment of Melasma.

Study design: Randomized-controlled trial (RCT). Study setting and duration: Dept of dermatology, CMH-Abbottabad, Nov-2022 /April-2023.

Methodology: The sample size of 60 patients 20 to 40 years were calculated by using Openepi App. The informed consent was taken. The patients were randomly allocated to two groups: Group A (30 patients injected with Intradermal Tranexamic acid (4mg/ml) and Group B (30 patients treated with PRP (1ml) intra-dermally, every fourth week for up to 12 weeks between both groups). The mMASI scale was used to evaluate all patients. The final evaluation was performed on the 24th week of follow-up. For analysis Statistical Package for the social sciences version-27 was used. To determine statistical significance a paired t-samples test with a p-value of < 0.05 was applied.

ELIGIBILITY:
Inclusion Criteria:

* 20_40 years of age
* suffering from melasma

Exclusion Criteria:

* pregnancy
* breastfeeding mothers
* allergic to tranexamic acid
* bleeding disorders
* warts or facial eczema

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Melasma severity index | 24 weeks
  Modified melasma area severity score is used to measure effectiveness of both drugs in treatment of melasma Score value ranges from 0-24 . 24 means melasma is more severe

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Dr sana aslam, Abbottabad, Khyber Pakhtun Khwaa
  - Sana aslam, Abbottabad, Khyber Pakhtun Khwa
  - Sana aslam, Abbottābād, Khyber Pakhtun Khwa